CLINICAL TRIAL: NCT01014039
Title: Telemark Polyp Study, a Randomized Trial on Colonoscopy Screening
Brief Title: Telemark Polyp Study, a Trial on Colonoscopy Screening
Acronym: TPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Department of Health and Social Affairs (Other Government)
Responsible Party: Principal Investigator, Geir Hoff, Professor, Norwegian Department of Health and Social Affairs
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TPS
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flexible Sigmoidoscopy Screening arm (Active Comparator): Intervention by flexible sigmoidoscopy screening
  Interventions: Procedure: Flexible Sigmoidoscopy Screening arm
- Control arm (No Intervention): No intervention (no screening)

INTERVENTIONS:
Procedure: Flexible Sigmoidoscopy Screening arm — sigmoidoscopy screening
  Other Names: polypectomy
  Arms: Flexible Sigmoidoscopy Screening arm

SUMMARY:
Colonoscopy screening to reduce mortality and incidence of colorectal cancer (CRC) has been implemented in many western countries. The estimated effect is based on case-control and observational studies. There are no randomized trials quantifying the effect of colonoscopy screening on CRC incidence and mortality.

The present study investigates the effect of a population-based once-only colonoscopy screening with polypectomy on the incidence of CRC in an average risk population.

In 1983, 900 individuals 55 to 64 years of age were randomly drawn from the population registry of Telemark county, Norway. 400 of these were invited to a flexible sigmoidoscopy screening examination, and 400 individuals were not offered any screening. In 1996, the remainder, both cohorts from 1983 were invited to a colonoscopy screening examination. A new age and sex matched control group, not being offered screening, was randomly drawn from the same registry. Both groups are to be followed with regard to CRC incidence, CRC mortality and all-cause mortality through national Norwegian registries.

DETAILED DESCRIPTION:
This as a randomized study of once-only colonoscopy screening (n=685) vs/no screening(care as usual)(n=684). Men and women at 63-72 years of age are recruited from the population registry. The intervention group is invited for screening after a bowel cleansing regimen at home. Follow-up is restricted to trace events (colorectal cancer incidence and deaths) through national registries.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 to 64 years old
* Both male and female

Exclusion criteria:

- Colorectal cancer diagnosed before study entry

Ages: 55 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1433 (Actual)
Dates: Start 1983-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Colorectal cancer mortality | at least 15 years of follow-up

SECONDARY OUTCOMES:
All cause mortality | at least 15 years of follow-up
colorectal cancer incidence | at least 15 years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Geir Hoff, MD, Study Chair — Sykehuset Telemark
Locations (1):
- Cancer Registry of Norway, Oslo, Norway